CLINICAL TRIAL: NCT02273271
Title: Evaluation of 3'-Deoxy-3'-[18F]Fluorothymidine -PET and Diffusion Weighted Imaging -MRI in Patients With Early Stage Non-small Cell Lung Cancer Treated With a Platinum-based Doublet as Preoperative Chemotherapy
Brief Title: Evaluation of FLT-PET and DWI-MRI in Patients With NSCLC Treated With a Platinum-based Doublet as Preoperative Chemo
Acronym: EVIDENCE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: European Organisation for Research and Treatment of Cancer - EORTC (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: EORTC-1217
Record Dates: First submitted 2014-10-16; First posted 2014-10-23 (Estimated); Last update posted 2015-10-30 (Estimated); Status verified 2015-10

CONDITIONS: Non-small Cell Lung Carcinoma
Keywords: FLT-PET; DWI-MRI
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Imaging arm (Experimental): 18F-FLT-PET/CT and DWI-MRI scans at baseline, at 14 days after first administration of chemotherapy and after up to 4 cycles of chemotherapy
  Interventions: Other: 18F-FLT-PET/CT and DWI-MRI

INTERVENTIONS:
Other: 18F-FLT-PET/CT and DWI-MRI — Patients with NSCLC will undergo 18F-FLT-PET/CT and DWI-MRI scans on three separate occasions. Dedicated in-house developed software will be used to quantify 18F-FLT SUV and ADC to assess tumor characteristics and response to therapy.

SUMMARY:
The purpose of the study is to qualify, independently, tumor cell proliferation by 3'-Deoxy-3'-[18F]Fluorothymidine (FLT) -Positron Emission Tomography , and cell death by Diffusion Weighted Imaging (DWI) -Magnetic Resonance Imaging (MRI) compared to pathological quantification (% of viable tumor cells) of the primary tumor after pre-operative chemotherapy in patients with operable Non Small Cell Lung Cancer (NSCLC).

DETAILED DESCRIPTION:
This is a prospective, multicenter, single-arm imaging trial. Patients with NSCLC will undergo 18F-FLT-PET/CT and DWI-MRI scans on three separate occasions: at baseline, at 14 days (maximum +/- 1 days deviation is acceptable) after first administration of chemotherapy and finally after up to 4 cycles of chemotherapy, and then followed by surgery. The quantification of 18F-FLT SUV and ADC will be measured to assess tumor characteristics and response to therapy.

Patients will be first registered into the EORTC system after signing the informed consent form. The site will have to complete all the study related procedures within 6 weeks prior to treatment and all eligibility criteria should be met before the patient can be enrolled into the study.

Both 18F-FLT-PET/CT and DWI-MRI will be assessed independently in this trial. Therefore the overall type I error of 0.1 will be split by two in order to test independently each imaging biomarker with a one-sided type I error of 0.05. In order to demonstrate with 95% confidence interval (one sided) that the correlation between the imaging biomarker change and the pathological response is > 0.5 (H0: rho ≤ 0.5) with 90% power if the true correlation is 0.8 (H1: rho > 0.5), 31 lesions are needed. As, in this population, patients only have the primary tumor, 31 eligible and evaluable patients will be needed for each primary endpoint.

If all included patients have both 18F-FLT-PET/CT and DWI-MRI then 31 eligible and evaluable patients will be enough. If some patients have only one type of scans (18F-FLT-PET/CT or DWI-MRI), the sample size would need to be adapted to have 31 patients with each type of scans.

In addition, the total number of patients to be registered may be increased to 40 patients for each primary endpoint to take into account some screening failure.

For the primary analysis of correlation between relative change in imaging biomarkers (18F-FLT-SUV or ADC) and pathological quantification, the correlation coefficient will be reported using a one-sided 95% confidence interval, and tested as a one-sided comparison to the null hypothesis (H0: ρ ≤ 0.5). All secondary objectives to correlate preoperative imaging biomarkers and IHC biological markers or tumor volume will use the same analysis as cited above with 99% confidence intervals. All measures will be analyzed in a random effect ANOVA model allowing for within center-variability.

Quality assurance is planned for the control of data consistency, on-site monitoring, audits, and quality assurance in pathological response assessment and in imaging.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* WHO performance status 0-1 (Appendix C)
* Histologically or cytological confirmed clinical stage II-IIIA non-small cell lung carcinoma (NSCLC), according to 7th TNM classification (Appendix D) (NOTE: patients with resectable N2 disease are also eligible)
* Baseline standard imaging assessment & staging should be performed within 6 weeks prior to planned treatment start.
* Patients must be candidate for curative intent surgery, and must be expected to complete the treatment.

  ♦♦ Adequate hematology and biochemical investigations, (should be done maximum 6 weeks before treatment starts)
* Normal bone marrow function based on routine blood samples, i.e. neutrophils ≥ 1.5 x 109/L, platelets ≥ 75 x 109/L, hemoglobin ≥ 10.0 g/dL
* Normal kidney function creatinine clearance ≥ 60 mL/min,
* Normal liver function assessed by routine laboratory examinations, i.e. bilirubin < 1.5 x upper limit of normal (ULN), ALT< 3 x ULN
* Patients must not have any contraindication for 18F-FLT-PET/CT or MRI procedures.
* Patient primary lung tumor larger than 20 mm in diameter (measured by diagnostic CT or MRI).
* Women of child bearing potential (WOCBP) must have a negative serum (or urine) pregnancy test before trial registration.
* Patients of childbearing / reproductive potential should use adequate birth control measures, as defined by the investigator, during the study treatment period and for at least 6 months after the last study procedure. A highly effective method of birth control is defined as those which result in low failure rate (i.e. less than 1% per year) when used consistently and correctly.
* Female subjects who are breast feeding should discontinue nursing before trial registration.
* Before patient registration, written informed consent must be given according to ICH/GCP, and national/local regulations.

Exclusion Criteria:

* Prior or current anticancer treatment for NSCLC, pre-operative therapy will include only chemotherapeutic drugs (pemetrexed is contraindicated), no other biological, targeted or radiotherapy is allowed
* Treatment with any investigational drug substance within 4 weeks prior to registration.
* Other malignancies in the 3 years prior to study entry with the exception of surgically cured carcinoma in situ of the cervix, in situ breast cancer, incidental finding of stage T1a or T1b prostate cancer, and basal/squamous cell carcinoma of the skin
* Evidence of any medical condition which would impair the ability of the patient to participate in the trial or might preclude therapy with chemotherapeutic drugs according to routine medical practice (e.g. unstable or uncompensated respiratory, cardiac, hepatic or renal disease, known dihydropyrimidine dehydrogenase deficiency, active infection, uncontrolled diabetes mellitus; uncontrolled arterial hypertension, history of unstable myocardial infarction)
* Any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule; those conditions should be discussed with the patient before randomization in the trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Estimated)
Dates: Start 2015-10; Primary Completion 2016-12 (Estimated); Study Completion 2017-02 (Estimated)

PRIMARY OUTCOMES:
Percentage of Apparent Diffusion Coefficient (ADC) change | day 14 relative to baseline
  Percentage of Apparent Diffusion Coefficient (ADC) change at day 14 relative to baseline
Percentage of FLT uptake change | day 14 relative to baseline
  Percentage of FLT uptake change at day 14 relative to baseline
Pathological quantification (% viable residual tumor cells) | in average at week 16 from baseline
  participants will receive chemotherapy for up to 12 weeks (4 cycles) and followed by surgery (with an expected surgical preparation of 2-4 weeks)

SECONDARY OUTCOMES:
Pre-operative (post-treatment) ADC measurement | in average at week 15 from baseline
  participants will receive chemotherapy for up to 12 weeks (4 cycles) and performed the DWI-MRI scan within one week prior to the surgery
Pre-operative (post-treatment) FLT uptake measurement | in average at week 15 from baseline
  participants will receive chemotherapy for up to 12 weeks (4 cycles) and performed the FLT-PET scan within one week prior to the surgery
Tumor volume (baseline, day 14 and post-treatment) | baseline, day 14 and post-treatment
Immunohistochemistry (IHC) cell proliferation marker Ki-67 | 1y
  Immunohistochemistry (IHC) cell proliferation marker Ki-67-index in diagnostic biopsy samples (if available) and surgical specimens.
Metabolic change from FDG-PET (if available) | in average at week 9 from baseline
  standard imaging per routine practice

CONTACTS AND LOCATIONS:
Overall Officials: Nandita deSouza, Principal Investigator — Royal Marsden Hospital - Sutton, Surrey; Sanjay Popat, Study Chair — Royal Marsden Hospital - Chelsea, London
Locations (2):
- Istituto Clinico Humanitas, Milan, Italy
- Royal Marsden Hospital - Sutton, Surrey, Sutton, United Kingdom